CLINICAL TRIAL: NCT03480360
Title: Haploidentical Allogeneic Peripheral Blood Transplantation: Clinical Trial and Laboratory Correlates Examining Checkpoint Immune Regulators' Expression
Brief Title: Haploidentical Allogeneic Peripheral Blood Transplantation: Examining Checkpoint Immune Regulators' Expression
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Kenneth Meehan, Principal Investogator- Kenneth Meehan, MD Staff Physician, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D17170
Record Dates: First submitted 2018-01-08; First posted 2018-03-29 (Actual); Results first posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-06

CONDITIONS: Acute Myeloid Leukemia; Chronic Lymphocytic Leukemia; Chronic Myeloid Leukemia; Myelodysplasia; Myeloproliferative Disorder; Myelofibrosis; Lymphoma; Lymphoma, Non-Hodgkin; Plasma Cell Disorder
Keywords: haploidentical; transplant; peripheral blood; allogeneic
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Anemia, Refractory, with Excess of Blasts; Myeloproliferative Disorders; Primary Myelofibrosis; Lymphoma; Lymphoma, Non-Hodgkin; Neoplasms, Plasma Cell | interventions — Cyclophosphamide; fludarabine; Whole-Body Irradiation; Tacrolimus; Mycophenolic Acid; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Johns Hopkins' conditioning regimen (Other): Cyclophosphamide, fludarabine, total body irradiation, immune suppression including tacrolimus and cellcept, Granulocyte colony-stimulating factor (G-CSF), and peripheral blood transplant
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Radiation: Total Body Irradiation; Drug: Tacrolimus; Drug: cellcept; Drug: g-csf; Procedure: Peripheral Blood Transplant

INTERVENTIONS:
Drug: Cyclophosphamide — 14.5 mg/kg for 2 days (days -6, -5) and then 50 mg/kg for two days (days 3, 4)
Drug: Fludarabine — 30 mg/m2 daily for 5 days
Radiation: Total Body Irradiation — 200 centigray (cGy) for one day (day -1)
Drug: Tacrolimus — 1 mg IV daily, (or the oral equivalent) adjusted to achieve a level between 5 and 15 ng/ml. If there is no evidence of GVHD, discontinue Tacrolimus by Day 180.
Drug: cellcept — dose at 15 mg/kg po three times per day (maximum dose of 3 grams/day). Stop Cellcept at Day 35 following transplantation.
Drug: g-csf — 5 mcg/kg/d starting day 5 and continue until Absolute Neutrophil Count (ANC) > 1000/mcL for 3 days.
Procedure: Peripheral Blood Transplant — cell dose goal: < 5 x 106 Hematopoietic progenitor cell antigen CD34+ cells/kg recipient weight

SUMMARY:
The standard Johns Hopkins' regimen will be used in study subjects, with the use of donor peripheral blood stem cells, rather than marrow. Clinical outcomes will be defined while focusing efforts on immune reconstitution focusing on immune checkpoint regulators after a related haploidentical stem cell transplant.

DETAILED DESCRIPTION:
We propose a clinical trial to define clinical endpoints, including engraftment, 100-day survival and one year survival (Objective #1). We will characterize the incidence, prevalence and function of immune checkpoint regulators in patients' blood and bone marrow following transplantation (Objective #2). We will correlate these laboratory results with clinical outcomes and the incidence of GVHD. As an exploratory aim, in those patients experiencing GVHD and requiring treatment, we will define the frequency/expression of checkpoint regulator expression and correlate these results with the patient's response to GVHD therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age: less than 75 years
* The patient must be approved for transplant by the treating transplant physician. This includes completion of their pre-transplant workup, as directed by standard Dartmouth-Hitchcock Medical Center (DHMC) Standard Operating Procedure (SOP) (DHMC SOP - Pre-transplant Evaluation of allogeneic recipient (Appendix).
* The patient must have a disease (listed below) with treatment-responsiveness that the treating transplant physician believes will benefit from an allogeneic stem cell transplant. The diseases include:
* Acute leukemia - Acute Myeloid Leukemia, Acute Lymphocytic Leukemia
* Chronic leukemia - Chronic Myeloid Leukemia, Chronic Lymphocytic Leukemia
* Myelodysplasia
* Myeloproliferative disorder
* Myelofibrosis
* Lymphoma - Non-Hodgkin's Lymphoma or Hodgkin's disease
* Plasma cell disorder, including myeloma, Waldenstrom's Macroglobulinemia
* Donor availability- the patient must have an identified RELATED haplo-identical donor
* No Human Immunodeficiency Virus infection or active hepatitis B or C
* Eastern Cooperative Oncology Group performance status: 0-2
* Diffusing capacity of carbon monoxide (DLCO) greater than or equal to 40 % predicted
* Left ventricular ejection fraction greater than or equal to 40%
* Serum bilirubin < 2x upper limit of normal; transaminases < 3x normal at the time of transplant
* No active or uncontrollable infection
* In female, a negative pregnancy test if experiencing menstrual periods
* No major organ dysfunction precluding transplantation
* No evidence of an active malignancy that would limit the patient's survival to less than 2 years. (If there is any question, the PI can make a decision).

Exclusion Criteria:

* Psychiatric disorder or a mental deficiency of the patient that is sufficiently severe to make compliance with the treatment unlikely, and making informed consent impossible.
* Major anticipated illness or organ failure incompatible with survival from bone marrow transplant.
* History of refractory systemic infection

DONOR ELIGIBILITY

* Human leukocyte antigen (HLA) haplo-identical matched related.
* The donor must be healthy and must be willing to serve as a donor, based on standard National Marrow Donor Program (NMDP) guidelines and DHMC SOP - Donor Evaluation (Appendix)
* The donor must have no significant co-morbidities that would put the donor at marked increased risk
* There is no age restriction for the donor
* Informed consent must be signed by donor

DONOR EXCLUSION CRITERIA

* The NMDP guidelines for exclusion criteria will be used (Appendix). In addition, the following donors are NOT eligible:
* Pregnant or lactating donor
* HIV or active Hep B or C in the donor
* Donor unfit to receive G-CSF and undergo apheresis
* A donor with a psychiatric disorder or mental deficiency that makes compliance with the procedure unlikely and informed consent impossible

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2025-09-13 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Meehan, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Norris Cotton Cancer Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bashey A, Zhang X, Sizemore CA, Manion K, Brown S, Holland HK, Morris LE, Solomon SR. T-cell-replete HLA-haploidentical hematopoietic transplantation for hematologic malignancies using post-transplantation cyclophosphamide results in outcomes equivalent to those of contemporaneous HLA-matched related and unrelated donor transplantation. J Clin Oncol. 2013 Apr 1;31(10):1310-6. doi: 10.1200/JCO.2012.44.3523. Epub 2013 Feb 19. PMID 23423745
- [Background] Solomon SR, Sizemore CA, Sanacore M, Zhang X, Brown S, Holland HK, Morris LE, Bashey A. Haploidentical transplantation using T cell replete peripheral blood stem cells and myeloablative conditioning in patients with high-risk hematologic malignancies who lack conventional donors is well tolerated and produces excellent relapse-free survival: results of a prospective phase II trial. Biol Blood Marrow Transplant. 2012 Dec;18(12):1859-66. doi: 10.1016/j.bbmt.2012.06.019. Epub 2012 Aug 1. PMID 22863841
- [Background] Ciurea SO, Zhang MJ, Bacigalupo AA, Bashey A, Appelbaum FR, Aljitawi OS, Armand P, Antin JH, Chen J, Devine SM, Fowler DH, Luznik L, Nakamura R, O'Donnell PV, Perales MA, Pingali SR, Porter DL, Riches MR, Ringden OT, Rocha V, Vij R, Weisdorf DJ, Champlin RE, Horowitz MM, Fuchs EJ, Eapen M. Haploidentical transplant with posttransplant cyclophosphamide vs matched unrelated donor transplant for acute myeloid leukemia. Blood. 2015 Aug 20;126(8):1033-40. doi: 10.1182/blood-2015-04-639831. Epub 2015 Jun 30. PMID 26130705
- [Background] Luznik L, O'Donnell PV, Symons HJ, Chen AR, Leffell MS, Zahurak M, Gooley TA, Piantadosi S, Kaup M, Ambinder RF, Huff CA, Matsui W, Bolanos-Meade J, Borrello I, Powell JD, Harrington E, Warnock S, Flowers M, Brodsky RA, Sandmaier BM, Storb RF, Jones RJ, Fuchs EJ. HLA-haploidentical bone marrow transplantation for hematologic malignancies using nonmyeloablative conditioning and high-dose, posttransplantation cyclophosphamide. Biol Blood Marrow Transplant. 2008 Jun;14(6):641-50. doi: 10.1016/j.bbmt.2008.03.005. PMID 18489989
- [Background] Mielcarek M, Martin PJ, Leisenring W, Flowers ME, Maloney DG, Sandmaier BM, Maris MB, Storb R. Graft-versus-host disease after nonmyeloablative versus conventional hematopoietic stem cell transplantation. Blood. 2003 Jul 15;102(2):756-62. doi: 10.1182/blood-2002-08-2628. Epub 2003 Mar 27. PMID 12663454
- [Background] Giralt S, Logan B, Rizzo D, Zhang MJ, Ballen K, Emmanouilides C, Nath R, Parker P, Porter D, Sandmaier B, Waller EK, Barker J, Pavletic S, Weisdorf D. Reduced-intensity conditioning for unrelated donor progenitor cell transplantation: long-term follow-up of the first 285 reported to the national marrow donor program. Biol Blood Marrow Transplant. 2007 Jul;13(7):844-52. doi: 10.1016/j.bbmt.2007.03.011. Epub 2007 May 24. PMID 17580263
- [Background] Kekre N, Antin JH. Hematopoietic stem cell transplantation donor sources in the 21st century: choosing the ideal donor when a perfect match does not exist. Blood. 2014 Jul 17;124(3):334-43. doi: 10.1182/blood-2014-02-514760. Epub 2014 Jun 9. PMID 24914138
- [Background] Bayraktar UD, Champlin RE, Ciurea SO. Progress in haploidentical stem cell transplantation. Biol Blood Marrow Transplant. 2012 Mar;18(3):372-80. doi: 10.1016/j.bbmt.2011.08.001. Epub 2011 Aug 9. PMID 21835146
- [Background] Parmesar K, Raj K. Haploidentical Stem Cell Transplantation in Adult Haematological Malignancies. Adv Hematol. 2016;2016:3905907. doi: 10.1155/2016/3905907. Epub 2016 May 30. PMID 27313619
- [Background] Luznik L, Engstrom LW, Iannone R, Fuchs EJ. Posttransplantation cyclophosphamide facilitates engraftment of major histocompatibility complex-identical allogeneic marrow in mice conditioned with low-dose total body irradiation. Biol Blood Marrow Transplant. 2002;8(3):131-8. doi: 10.1053/bbmt.2002.v8.pm11939602.
- [Background] Ciurea SO, Mulanovich V, Saliba RM, Bayraktar UD, Jiang Y, Bassett R, Wang SA, Konopleva M, Fernandez-Vina M, Montes N, Bosque D, Chen J, Rondon G, Alatrash G, Alousi A, Bashir Q, Korbling M, Qazilbash M, Parmar S, Shpall E, Nieto Y, Hosing C, Kebriaei P, Khouri I, Popat U, de Lima M, Champlin RE. Improved early outcomes using a T cell replete graft compared with T cell depleted haploidentical hematopoietic stem cell transplantation. Biol Blood Marrow Transplant. 2012 Dec;18(12):1835-44. doi: 10.1016/j.bbmt.2012.07.003. Epub 2012 Jul 11. PMID 22796535
- [Background] Chang YJ, Zhao XY, Huang XJ. Immune reconstitution after haploidentical hematopoietic stem cell transplantation. Biol Blood Marrow Transplant. 2014 Apr;20(4):440-9. doi: 10.1016/j.bbmt.2013.11.028. Epub 2013 Dec 4. PMID 24315844
- [Background] Habicht A, Kewalaramani R, Vu MD, Demirci G, Blazar BR, Sayegh MH, Li XC. Striking dichotomy of PD-L1 and PD-L2 pathways in regulating alloreactive CD4(+) and CD8(+) T cells in vivo. Am J Transplant. 2007 Dec;7(12):2683-92. doi: 10.1111/j.1600-6143.2007.01999.x. Epub 2007 Oct 9. PMID 17924994
- [Background] Schilbach K, Schick J, Wehrmann M, Wollny G, Simon P, Schlegel PG, Eyrich M. PD-1-PD-L1 pathway is involved in suppressing alloreactivity of heart infiltrating t cells during murine gvhd across minor histocompatibility antigen barriers. Transplantation. 2007 Jul 27;84(2):214-22. doi: 10.1097/01.tp.0000268074.77929.54. PMID 17667813
- [Background] Blazar BR, Taylor PA, Panoskaltsis-Mortari A, Sharpe AH, Vallera DA. Opposing roles of CD28:B7 and CTLA-4:B7 pathways in regulating in vivo alloresponses in murine recipients of MHC disparate T cells. J Immunol. 1999 Jun 1;162(11):6368-77. PMID 10352249
- [Background] Wallace PM, Johnson JS, MacMaster JF, Kennedy KA, Gladstone P, Linsley PS. CTLA4Ig treatment ameliorates the lethality of murine graft-versus-host disease across major histocompatibility complex barriers. Transplantation. 1994 Sep 15;58(5):602-10. doi: 10.1097/00007890-199409150-00013. PMID 8091487
- [Background] Al-Chaqmaqchi H, Sadeghi B, Abedi-Valugerdi M, Al-Hashmi S, Fares M, Kuiper R, Lundahl J, Hassan M, Moshfegh A. The role of programmed cell death ligand-1 (PD-L1/CD274) in the development of graft versus host disease. PLoS One. 2013 Apr 4;8(4):e60367. doi: 10.1371/journal.pone.0060367. Print 2013. PMID 23593203
- [Background] Le Mercier I, Chen W, Lines JL, Day M, Li J, Sergent P, Noelle RJ, Wang L. VISTA Regulates the Development of Protective Antitumor Immunity. Cancer Res. 2014 Apr 1;74(7):1933-44. doi: 10.1158/0008-5472.CAN-13-1506. PMID 24691994
- [Background] Lines JL, Sempere LF, Broughton T, Wang L, Noelle R. VISTA is a novel broad-spectrum negative checkpoint regulator for cancer immunotherapy. Cancer Immunol Res. 2014 Jun;2(6):510-7. doi: 10.1158/2326-6066.CIR-14-0072. PMID 24894088
- [Background] Liu J, Yuan Y, Chen W, Putra J, Suriawinata AA, Schenk AD, Miller HE, Guleria I, Barth RJ, Huang YH, Wang L. Immune-checkpoint proteins VISTA and PD-1 nonredundantly regulate murine T-cell responses. Proc Natl Acad Sci U S A. 2015 May 26;112(21):6682-7. doi: 10.1073/pnas.1420370112. Epub 2015 May 11. PMID 25964334
- [Background] Highfill SL, Rodriguez PC, Zhou Q, Goetz CA, Koehn BH, Veenstra R, Taylor PA, Panoskaltsis-Mortari A, Serody JS, Munn DH, Tolar J, Ochoa AC, Blazar BR. Bone marrow myeloid-derived suppressor cells (MDSCs) inhibit graft-versus-host disease (GVHD) via an arginase-1-dependent mechanism that is up-regulated by interleukin-13. Blood. 2010 Dec 16;116(25):5738-47. doi: 10.1182/blood-2010-06-287839. Epub 2010 Aug 31. PMID 20807889
- [Background] Messmann JJ, Reisser T, Leithauser F, Lutz MB, Debatin KM, Strauss G. In vitro-generated MDSCs prevent murine GVHD by inducing type 2 T cells without disabling antitumor cytotoxicity. Blood. 2015 Aug 27;126(9):1138-48. doi: 10.1182/blood-2015-01-624163. Epub 2015 Jul 16. PMID 26185131
- [Background] Rieber N, Wecker I, Neri D, Fuchs K, Schafer I, Brand A, Pfeiffer M, Lang P, Bethge W, Amon O, Handgretinger R, Hartl D. Extracorporeal photopheresis increases neutrophilic myeloid-derived suppressor cells in patients with GvHD. Bone Marrow Transplant. 2014 Apr;49(4):545-52. doi: 10.1038/bmt.2013.236. Epub 2014 Jan 27. PMID 24464140

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 21 individuals signed consent. 1 individual was deemed ineligible during screening. Therefore 20 individuals were evaluated for the primary endpoint.
Period: Overall Study
Arm/Group | Johns Hopkins' Conditioning Regimen
Started | 20
Completed | 18
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | Johns Hopkins' Conditioning Regimen
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 9
  >=65 years | 10
Age, Continuous [Mean (Full Range); unit: Years] | 59.55 [18 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20
Number of Evaluable Participants [Number; unit: participants] | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Survived to 100-Days Post-transplant
Description: Define 100-day survival of subjects
Time Frame: 100 days post date of peripheral blood transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Johns Hopkins' Conditioning Regimen
Number analyzed (Participants) | 20
Participants | 18

2. Primary Outcome: Number of Participants Who Survived to One Year Post-Transplant.
Description: Define one year survival of subjects
Time Frame: One year post date of peripheral blood transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Johns Hopkins' Conditioning Regimen
Number analyzed (Participants) | 20
Participants | 16

3. Primary Outcome: Number of Participants Who Experienced a Successful Engraftment
Description: Define number of subjects who experience a successful engraftment: Defined as absolute neutrophil count > 500/mm3 and platelets > 20,000/mcl for three consecutive days (count first day as engraftment)
Time Frame: Post-peripheral blood transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Johns Hopkins' Conditioning Regimen
Number analyzed (Participants) | 20
Participants | 18

4. Primary Outcome: Number of Participants Who Achieved a Response to Treatment at 100 Days
Description: Define response to treatment at 100 days post-peripheral blood transplant. The Standard International Criteria for responses for each disease will be used, based on CIBMTR (Center for International Blood and Marrow Transplant Research) criteria.
Time Frame: 100 days post-peripheral blood transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Johns Hopkins' Conditioning Regimen
Number analyzed (Participants) | 20
Participants | 16

5. Primary Outcome: Number of Participants Who Achieved a Response to Treatment at One Year
Description: Define response to treatment at one year post-peripheral blood transplant. The Standard International Criteria for responses for each disease will be used, based on CIBMTR (Center for International Blood and Marrow Transplant Research) criteria.
Time Frame: One year post-peripheral blood transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Johns Hopkins' Conditioning Regimen
Number analyzed (Participants) | 20
Participants | 13

6. Primary Outcome: Number of Participants Who Experienced Toxicities Associated With This Treatment Regimen
Description: Define subjects who experienced toxicities associated with this treatment regimen
Time Frame: Post-peripheral blood transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Johns Hopkins' Conditioning Regimen
Number analyzed (Participants) | 20
Participants | 16

7. Primary Outcome: Number of Participants Who Had Incidence of Acute GVHD
Description: Define subjects who had incidence of acute GVHD
Time Frame: Post-peripheral blood transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Johns Hopkins' Conditioning Regimen
Number analyzed (Participants) | 20
Participants | 3

8. Primary Outcome: Number of Participants Who Had Incidence of Chronic GVHD
Description: Define subjects who had incidence of chronic GVHD
Time Frame: Post-peripheral blood transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Johns Hopkins' Conditioning Regimen
Number analyzed (Participants) | 20
Participants | 9

9. Primary Outcome: Number of Participants Who Experienced Donor-Recipient Chimerism Following Transplant at Days 30, 60, and 90.
Description: Define subjects who experience donor-recipient chimerism following transplant at days 30, 60 and 90. All patients were assessed for donor-recipient chimerism at days 30, 60, and 90, but only one patient experienced chimerism. Day 90 for this patient is reported.
Time Frame: Days 30, 60, and 90 post-peripheral blood transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Johns Hopkins' Conditioning Regimen
Number analyzed (Participants) | 20
Participants | 1

10. Primary Outcome: Number of Participants Who Experienced Treatment-Related Mortality Within the First 100 Days
Description: Define subjects who experienced treatment-related mortality within the first 100 days post-peripheral blood transplant
Time Frame: 100 days post-peripheral blood transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Johns Hopkins' Conditioning Regimen
Number analyzed (Participants) | 20
Participants | 2

11. Secondary Outcome: Immune Checkpoint Regulators - Incidence
Description: To characterize the incidence of immune checkpoint regulators (V-domain Ig Suppressor of T-cell Activation, cytotoxic T-lymphocyte-associated protein 4 [CTLA], Programmed cell death protein 1 [PD-1]) during early immune recovery following an allogeneic stem cell transplant.
Time Frame: Days 30, 60, and 90 post-transplant
Population: Blood samples were collected, however laboratory analysis was not performed due to lack of funding. There are no plans to potentially analyze the samples in the future, therefore these samples were not, and will not be, analyzed.
Arm/Group | Johns Hopkins' Conditioning Regimen
Number analyzed (Participants) | 0

12. Secondary Outcome: Myeloid-derived Suppressor Cells (MDSCs) After Graft vs. Host Disease (GVHD) Diagnosis - Checkpoint Regulator Expression
Description: In those patients experiencing GVHD, the study team will define the checkpoint regulator expression on MDSCs
Time Frame: Post-transplant through study completion or death, assessed up to 3 years post-transplant
Population: as for outcome 11
Arm/Group | Johns Hopkins' Conditioning Regimen
Number analyzed (Participants) | 0

13. Secondary Outcome: MDSCs After GVHD Diagnosis - Peripheral Blood Mononuclear Cells
Description: In those patients experiencing GVHD, the study team will define the peripheral blood mononuclear cells and myeloid subsets.
Time Frame: Post-transplant through study completion or death, assessed up to 3 years post-transplant
Population: as for outcome 11
Arm/Group | Johns Hopkins' Conditioning Regimen
Number analyzed (Participants) | 0

14. Secondary Outcome: MDSCs After GVHD Diagnosis - Myeloid Subsets Using Flow Cytometry
Description: In those patients experiencing GVHD, the study team will define the myeloid subsets.
Time Frame: Post-transplant through study completion or death, assessed up to 3 years post-transplant
Population: as for outcome 11
Arm/Group | Johns Hopkins' Conditioning Regimen
Number analyzed (Participants) | 0

15. Secondary Outcome: MDSCs After GVHD Diagnosis - Frequency
Description: In those patients experiencing GVHD, the study team will define the MDSCs frequency.
Time Frame: Post-transplant through study completion or death, assessed up to 3 years post-transplant
Population: as for outcome 11
Arm/Group | Johns Hopkins' Conditioning Regimen
Number analyzed (Participants) | 0

16. Secondary Outcome: Immune Checkpoint Regulators - Prevalence
Description: To characterize the prevalence of immune checkpoint regulators (VISTA, CTLA-4, PD-1) during early immune recovery following an allogeneic stem cell transplant.
Time Frame: Days 30, 60, and 90 post-transplant
Population: as for outcome 11
Arm/Group | Johns Hopkins' Conditioning Regimen
Number analyzed (Participants) | 0

17. Secondary Outcome: Immune Checkpoint Regulators - Function
Description: Flow cytometry will be used to characterize the function of immune checkpoint regulators (VISTA, CTLA-4, PD-1) during early immune recovery following an allogeneic stem cell transplant.
Time Frame: Days 30, 60, and 90 post-transplant
Population: as for outcome 11
Arm/Group | Johns Hopkins' Conditioning Regimen
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Monitoring of all acute toxicities (grade 3 or higher) occurred until the time of discharge (post-transplant). After discharge, until day 100, only serious toxicities (grade 4 or higher) were recorded. All-Cause Mortality was monitored from the time of transplant to three years post-transplant.
Arm/Group | Johns Hopkins' Conditioning Regimen
All-Cause Mortality (participants affected / at risk) | 5/20
Serious Adverse Events (participants affected / at risk) | 3/20
Other Adverse Events (participants affected / at risk) | 16/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Johns Hopkins' Conditioning Regimen (N=20)
Edema Limbs (General disorders) | 1 (1) — Probably related to pseudo-gout
GI GVHD (Gastrointestinal disorders) | 1 (1)
Liver GVHD (Hepatobiliary disorders) | 1 (1)
Skin GVHD (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Johns Hopkins' Conditioning Regimen (N=20)
Anorexia (Blood and lymphatic system disorders) | 15 (18)
Edema (General disorders) | 4 (4)
Rigors (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Dysrhythmia (Cardiac disorders) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 5 (5)
C. Diff (Infections and infestations) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Delirium (Psychiatric disorders) | 2 (3)
Dysesthesia (Nervous system disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Central Line (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-04): https://cdn.clinicaltrials.gov/large-docs/60/NCT03480360/Prot_SAP_000.pdf